CLINICAL TRIAL: NCT00001012
Title: An Open Label, Multiple Dose Ranging Trial of AL721 in Patients With Persistent Generalized Lymphadenopathy and Symptomatic HIV Infection
Brief Title: A Study of AL721 in HIV-Infected Patients With Swollen Lymph Nodes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 022
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; T-Lymphocytes; Dose-Response Relationship, Drug; Drug Evaluation; Acquired Immunodeficiency Syndrome; AL 721; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — neutral lipid, phosphatidylcholine, phosphatidylethanolamine drug combination

INTERVENTIONS:
Drug: AL 721

SUMMARY:
To study the tolerance and safety of increasing doses of AL-721 in patients with persistent generalized lymphadenopathy (PGL) and symptomatic HIV infection, and to obtain preliminary information on the effectiveness of AL-721 against the human immunodeficiency virus (HIV) in HIV-infected persons with PGL and symptomatic HIV infection. Although zidovudine (AZT) prolongs life in certain AIDS patients, it is not a cure for AIDS and it also has toxic effects in many patients. Therefore, it is necessary to test other drugs in HIV-infected patients. AL-721 is a mixture of lipids (fats) extracted from egg yolks. Laboratory tests suggest that it might inhibit the infectivity of the HIV. AL-721 has been tried so far in a few patients for short periods of time and has been found to be well tolerated.

DETAILED DESCRIPTION:
Although zidovudine (AZT) prolongs life in certain AIDS patients, it is not a cure for AIDS and it also has toxic effects in many patients. Therefore, it is necessary to test other drugs in HIV-infected patients. AL-721 is a mixture of lipids (fats) extracted from egg yolks. Laboratory tests suggest that it might inhibit the infectivity of the HIV. AL-721 has been tried so far in a few patients for short periods of time and has been found to be well tolerated.

Patients receive AL-721 twice daily. The first dose is taken on an empty stomach 1 hour before a fat-free breakfast, with specific instructions given on foods that are allowed; the second dose is taken at least 3 hours after the evening meal. No snacks are permitted after the evening meal or after the evening dose of study medication. The study is scheduled to last for 16 weeks of treatment and 4 weeks of follow-up. Throughout the study, frequent blood samples will be taken from an arm vein. The blood samples are studied to evaluate any changes in the patient's immune system, any toxic effects that might be detected in the blood, and any changes in the presence of the HIV in the blood.

ELIGIBILITY:
Inclusion Criteria

* Persistent generalized lymphadenopathy (PGL) (CDC-Group III), defined as palpable lymphadenopathy (nodes of 1 cm or greater) at two or more noncontiguous extrainguinal sites persisting for > 3 months in the absence of an illness other than HIV infection to account for the findings.
* AIDS related complex (ARC), defined as the presence of at least one of the following findings within 12 months prior to entry and the absence of a concurrent illness or condition other than HIV infection to explain the findings:
* Any findings which define CDC-Group IV A.
* History of any one of the findings that define CDC-Group IV C2.
* Patients with any of the ARC symptoms can also have PGL and be enrolled in the protocol as ARC patients.
* A positive antibody to HIV by any federally licensed ELISA test kit within 30 days of entry.

Concurrent Medication: Allowed:

* Topical or oral antifungal, antiviral, or antibiotic agents to treat oral candidiasis, herpes simplex, herpes zoster, or bacterial infections that develop during the course of the study.

Exclusion Criteria

* Exclude hemophiliacs.
* Active substance abuse.
* Alcohol consumption should be kept to a minimum.

Co-existing Condition:

Patients with the following will be excluded:

* Hemophilia.
* History or presence of an AIDS-defining opportunistic infection or malignancy.
* AIDS related complex (ARC) patients with prior (within the last 12 months) or current history of diarrhea defined as = or > 3 liquid stools per day persisting for longer than 1 month.
* Significant malabsorption:
* Greater than 10 percent weight loss within past 3 months with serum carotene < 75 IU/ml or vitamin A < 75 IU/ml.
* Significant cardiac, liver, renal, or neurologic disorder.
* Active ARC-defining secondary infection (oral candidiasis, oral hairy leukoplakia, multidermatomal herpes zoster, recurrent nontyphoidal Salmonella bacteremia or Nocardiosis) undergoing therapy or prophylaxis within 7 days of study entry.
* Active tuberculosis under treatment.
* Concurrent neoplasm other than basal cell carcinoma of the skin or in situ carcinoma of the cervix.

Concurrent Medication:

Excluded:

* Any medication that will interfere with the assessment of AL-721, including nutritional supplements, vitamins, laxatives, and over-the-counter products containing lecithin.
* Chemoprophylaxis for Pneumocystis carinii (PCP), candida, herpes simplex, herpes zoster infections, or bacterial infections.
* Intravenous topical or oral antifungal, antiviral, or antibiotic agents to treat oral candidiasis, herpes simplex, herpes zoster, or bacterial infections that develop during the course of the study.
* Systemic chemotherapy.

Prior Medication:

Excluded within 30 days of study entry:

* Any investigational drug.
* Biologic response modifiers.
* Corticosteroids.
* Chemotherapeutic agents.
* Excluded within 90 days of study entry:
* Any antiretroviral agent or AL-721.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50

CONTACTS AND LOCATIONS:
Overall Officials: Mildvan D, Study Chair; Armstrong D, Study Chair
Locations (9):
- United States (9):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Univ of Minnesota, Minneapolis, Minnesota
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York

REFERENCES:
- [Background] Mildvan D, Buzas J, Armstrong D, Antoniskis D, Sacks HS, Rhame FS, Mosbach EW, Pettinelli C. An open-label, dose-ranging trial of AL 721 in patients with persistent generalized lymphadenopathy and AIDS-related complex. J Acquir Immune Defic Syndr (1988). 1991;4(10):945-51. PMID 1890604